CLINICAL TRIAL: NCT07147543
Title: Study to Verify the Effectiveness and Safety of the Electrically Powered Orthopedic Exercise Device on Gait Ability in Patients With Gait Disorders : Investigator-Initiated, Single-Center, Single-Group Clinical Trial
Brief Title: Effectiveness and Safety of Electrically Powered Orthopedic Exercise Device for Gait Disorders
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9-2025-0021
Record Dates: First submitted 2025-04-21; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Gait Disorders
Keywords: Rehabilitation; Gait; Wearable robot; Gait Disorders
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Researchers will compare non-wearing and wearing conditions of the electrically powered orthopedic exercise device walking speeds, spatiotemporal parameters, balance, and satisfaction survey in participants and does not establish a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wearing conditions of Electrically Powered Orthopedic Exercise Device (Experimental): Participants will undergo gait and balance function tests under both non-wearing and wearing conditions of the electrically powered orthopedic exercise device
  Interventions: Device: Electrically Powered Orthopedic Exercise Device

INTERVENTIONS:
Device: Electrically Powered Orthopedic Exercise Device — Participants who pass the screening undergo an evaluation of gait function and balance ability without wearing the Electrically Powered Orthopedic Exercise Device. Afterward, the patient wears the motorized orthopedic exercise device for a total of four adaptation sessions. In each session, the patient performs short-distance walking within 10 meters while wearing the device to explore the appropriate assistive mode and level of support that match their physical condition. No evaluations are conducted while wearing the device during sessions 1, 2, and 3. After the 4th session, an evaluation identical to the one conducted without the device is performed while wearing it, and a satisfaction survey is conducted.

SUMMARY:
Aging is a global trend, and consequently, the prevalence of age-related diseases is increasing. Gait disorders are common among the elderly and can result not only from various underlying conditions affecting gait but also from the decline in physiological and neurological functions associated with the normal aging process.

Gait is a fundamental daily activity that requires the coordinated integration of the central and peripheral nervous systems, as well as the musculoskeletal system. Therefore, impairments in any of these systems-including the nervous, cardiovascular, respiratory, or musculoskeletal systems-can lead to gait dysfunction. Gait disorders negatively impact quality of life by increasing the risk of falls, reducing the ability to perform activities of daily living (ADLs), and limiting physical activity. Accordingly, various approaches to maintaining and improving gait function in older adults are being actively explored.

Currently, gait aids such as canes and walkers are commonly used to support individuals with gait impairments. These devices help redistribute body weight by providing a broader base of support, thereby assisting with balance and stability. However, they do not directly facilitate the movement of the lower limbs. To enhance gait function, numerous studies have investigated repetitive lower-limb movement training using bicycles or robotic devices. However, the extent of functional improvement resulting from such training remains unclear, and the long-term efficacy is still uncertain.

Recent advancements in sensing technology for joint motion and actuator efficiency have led to the development of wearable assistive devices that are significantly more compact and lightweight compared to conventional robotic systems. This study aims to evaluate the effectiveness of a newly developed electrically powered orthopedic exercise device in patients with gait disorders by assessing changes in gait parameters upon wearing the device, thereby exploring its clinical feasibility.

DETAILED DESCRIPTION:
(1) Overview of study design This investigator-initiated exploratory study is a pilot study designed to evaluate the effectiveness and safety of the Electrically Powered Orthopedic Exercise Device by measuring and analyzing gait function and balance ability in patients with gait disorders under both non-wearing and wearing conditions.

(2) Experimental Group and Evaluation Procedures

1. Participant Selection:

   This study includes a single test group with a total of 30 participants. The selection of participants for the electrically powered orthopedic exercise device and the overall study process will be conducted under the prescription and guidance of a rehabilitation medicine specialist, and supervised by assistants (physicians and occupational therapists). The examiner will collect clinical information and conduct a screening assessment for each participant.
2. Evaluation Phase Without Device:

   After the screening test, participants undergo assessments of walking ability and balance without wearing the motorized orthopedic exercise device. A 10-minute rest period is provided between each assessment. If the participant wishes, additional rest time is allowed and recorded in the case report form. The assessments include the 10-Meter Walk Test, the 6-Minute Walk Test, the Timed Up and Go Test, and the Berg Balance Scale. These evaluations are conducted in the rehabilitation function testing room on the second floor of the facility under the supervision of the research team (physician and either a physical or occupational therapist).
3. Pre-Adaptation Phase:

   After the evaluations without the device, a total of four adaptation sessions are conducted, during which the participant wears the device and performs short-distance walking within 10 meters. These sessions are designed to help the participant become familiar with the operation and wearing method of the H10 device. Appropriate device settings are configured for each participant to minimize any potential inexperience or anxiety during use. Participants must complete all four adaptation sessions, and each session should be conducted within a two-week interval.
4. Evaluation Phase:

After completing all four adaptation sessions, participants undergo assessments of walking ability and balance while wearing the motorized orthopedic exercise device. A 10-minute rest period is provided between each assessment. If the participant wishes, additional rest time is allowed and recorded in the case report form. The assessments include the 10-Meter Walk Test, the 6-Minute Walk Test, the Timed Up and Go Test, and the Berg Balance Scale. These evaluations are conducted in the rehabilitation function testing room on the second floor of the facility under the supervision of the research team (physician and either a physical or occupational therapist). After the evaluations are completed, a usability and satisfaction survey regarding the motorized orthopedic exercise device is conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years or older
2. Patients experiencing subjective gait or balance disorders
3. Individuals who visited Yongin Severance Hospital, understood the study, voluntarily agreed to participate, and signed the consent form
4. Patients with a Functional Ambulatory Category (FAC) score of less than 4
5. Individuals who can sit on the edge of a bed without assistance and stand for 10 seconds with or without support
6. Individuals with sufficient cognitive ability to follow and understand simple instructions (Mini-Mental State Examination score ≥ 20)

Exclusion Criteria:

1. Individuals with contraindications to weight-bearing in the lower extremities, such as severe lower extremity joint contractures, osteoporosis, or untreated fractures
2. Individuals who cannot wear the device due to skin diseases or open wounds
3. Individuals with a significant discrepancy in lower extremity length
4. Individuals with severe lower extremity deformities or joint contractures
5. Individuals unable to maintain a sitting or standing posture independently
6. Individuals with severe cognitive impairment (Mini-Mental State Examination score < 20), delirium, or severe speech impairment preventing cooperation in wearing the device
7. Individuals unable to stand or walk for extended periods due to underlying conditions such as orthostatic hypotension or reduced cardiopulmonary function
8. Pregnant or potentially pregnant individuals
9. Individuals with other clinically significant conditions deemed inappropriate for this study by the principal investigator or research team based on medical judgment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-04-06 (Estimated); Study Completion 2026-04-06 (Estimated)

PRIMARY OUTCOMES:
10-Meter Walk Test | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  Patients are instructed to walk 14 m, including 2 m at both ends for acceleration and deceleration, at their comfortable speed. Gait speed was calculated by dividing the 10m distance by the time taken.

SECONDARY OUTCOMES:
Timed Up and Go (TUG) Test | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  Researchers ask patients to rise from a seated position, walk a distance of 3 m, turn around, return to the chair, and sit back. The average time of three trials was recorded as a result
6-Minute Walk Test | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  Patients are instructed to walk back and forth along the 30-meter path as many times as possible within 6 minutes. The examiner records the total distance covered, abnormal gait patterns, and the time of occurrence of any gait deviations.
Berg balance scale (BBS) | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  Patients are asked to perform 14 tasks regarding the static and dynamic balance of patients. Each task was rated on a five-point scale from 0 to 4, with a total score of 56.
Spatiotemporal Parameters of Gait : Total Step Count | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  While the participant performs the test wearing an insole-type gait analyzer, spatiotemporal gait parameters are collected and recorded.
  Total Step Count: The total number of steps taken during walking.
Spatiotemporal Parameters of Gait : Cadence | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  While the participant performs the test wearing an insole-type gait analyzer, spatiotemporal gait parameters are collected and recorded.
  Cadence: The number of steps taken per minute, measured in steps per minute (spm).
Spatiotemporal Parameters of Gait : Self-Selected Walking Speed | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  While the participant performs the test wearing an insole-type gait analyzer, spatiotemporal gait parameters are collected and recorded.
  Self-Selected Walking Speed: The participant's walking speed when walking naturally at a comfortable pace.
Spatiotemporal Parameters of Gait : Distance | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  While the participant performs the test wearing an insole-type gait analyzer, spatiotemporal gait parameters are collected and recorded.
  Distance: The total distance covered during walking, measured in meters (m).
Spatiotemporal Parameters of Gait : Stride Length | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  While the participant performs the test wearing an insole-type gait analyzer, spatiotemporal gait parameters are collected and recorded.
  Stride Length: The distance between the heel of one foot to the heel of the same foot during consecutive steps. Measured in meters (m), stride length is adjusted for height to account for differences in body size.
Satisfaction evaluation | Upon completion of the end-point assessment conducted on the same day as session 4
  Participants will complete a satisfaction survey for usability and satisfaction assessment of the electrically powered orthopedic exercise device, based on the Korean version of the Quebec User Evaluation of Satisfaction with assistive Technology (K-QUEST 2.0).21 This survey consists of 12 items on a 5-point scale. Participants rate their satisfaction with the assistive device and related services.
  (An average score of 4 or higher will be interpreted as positive satisfaction, an average score of 2 or lower will be interpreted as negative satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Na Young Kim, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Yongin Severance Hospital, Yongin-si, Gyeonggi-do, South Korea, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perera S, Mody SH, Woodman RC, Studenski SA. Meaningful change and responsiveness in common physical performance measures in older adults. J Am Geriatr Soc. 2006 May;54(5):743-9. doi: 10.1111/j.1532-5415.2006.00701.x. PMID 16696738
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Lee, Sang-Heon, Bong-Keun Jung, and So-Yeon Park. "Korean Translation and Psychometric Properties of Quebec User Evaluation of Satisfaction Assistive Technology 2.0." Journal of the Korea Academia-Industrial Cooperation Society. The Korea Academia-Industrial Cooperation Society, July 31, 2013.
- [Background] Bang DH, Shin WS. Effects of robot-assisted gait training on spatiotemporal gait parameters and balance in patients with chronic stroke: A randomized controlled pilot trial. NeuroRehabilitation. 2016 Apr 6;38(4):343-9. doi: 10.3233/NRE-161325. PMID 27061162
- [Background] Godi M, Franchignoni F, Caligari M, Giordano A, Turcato AM, Nardone A. Comparison of reliability, validity, and responsiveness of the mini-BESTest and Berg Balance Scale in patients with balance disorders. Phys Ther. 2013 Feb;93(2):158-67. doi: 10.2522/ptj.20120171. Epub 2012 Sep 27. PMID 23023812
- [Background] Guyatt GH, Sullivan MJ, Thompson PJ, Fallen EL, Pugsley SO, Taylor DW, Berman LB. The 6-minute walk: a new measure of exercise capacity in patients with chronic heart failure. Can Med Assoc J. 1985 Apr 15;132(8):919-23. PMID 3978515
- [Background] Dolny DG, Collins MG, Wilson T, Germann ML, Davis HP. Validity of lower extremity strength and power utilizing a new closed chain dynamometer. Med Sci Sports Exerc. 2001 Jan;33(1):171-5. doi: 10.1097/00005768-200101000-00026. PMID 11194105
- [Background] Kim Heon-tae, Moon Jun-bae, Ryu Seung-ho, and Kang Min-soo. Validity study of the Korean version of the International Physical Activity Questionnaire (IPAQ): Verification of construct-related validity. Korean Journal of Physical Education No. 2017;56
- [Background] Gajdosik RL, Bohannon RW. Clinical measurement of range of motion. Review of goniometry emphasizing reliability and validity. Phys Ther. 1987 Dec;67(12):1867-72. doi: 10.1093/ptj/67.12.1867. PMID 3685114
- [Background] Mehrholz J, Wagner K, Rutte K, Meissner D, Pohl M. Predictive validity and responsiveness of the functional ambulation category in hemiparetic patients after stroke. Arch Phys Med Rehabil. 2007 Oct;88(10):1314-9. doi: 10.1016/j.apmr.2007.06.764. PMID 17908575
- [Background] Cuthbert SC, Goodheart GJ Jr. On the reliability and validity of manual muscle testing: a literature review. Chiropr Osteopat. 2007 Mar 6;15:4. doi: 10.1186/1746-1340-15-4. PMID 17341308
- [Background] Kang Y, NA D-L, Hahn S. A validity study on the Korean Mini-Mental State Examination (K-MMSE) in dementia patients. Journal of the Korean neurological association 1997:300-308
- [Background] Tao Y, Luo J, Tian J, Peng S, Wang H, Cao J, Wen Z, Zhang X. The role of robot-assisted training on rehabilitation outcomes in Parkinson's disease: a systematic review and meta-analysis. Disabil Rehabil. 2024 Sep;46(18):4049-4067. doi: 10.1080/09638288.2023.2266178. Epub 2023 Oct 11. PMID 37818694
- [Background] Chou CH, Hwang CL, Wu YT. Effect of exercise on physical function, daily living activities, and quality of life in the frail older adults: a meta-analysis. Arch Phys Med Rehabil. 2012 Feb;93(2):237-44. doi: 10.1016/j.apmr.2011.08.042. PMID 22289232
- [Background] Sudarsky L. Gait disorders: prevalence, morbidity, and etiology. Adv Neurol. 2001;87:111-7. No abstract available. PMID 11347214
- [Background] Lange AK, Vanwanseele B, Fiatarone Singh MA. Strength training for treatment of osteoarthritis of the knee: a systematic review. Arthritis Rheum. 2008 Oct 15;59(10):1488-94. doi: 10.1002/art.24118. PMID 18821647
- [Background] Bennett DA, Beckett LA, Murray AM, Shannon KM, Goetz CG, Pilgrim DM, Evans DA. Prevalence of parkinsonian signs and associated mortality in a community population of older people. N Engl J Med. 1996 Jan 11;334(2):71-6. doi: 10.1056/NEJM199601113340202. PMID 8531961
- [Background] Salzman B. Gait and balance disorders in older adults. Am Fam Physician. 2010 Jul 1;82(1):61-8. PMID 20590073
- [Background] Mahlknecht P, Kiechl S, Bloem BR, Willeit J, Scherfler C, Gasperi A, Rungger G, Poewe W, Seppi K. Prevalence and burden of gait disorders in elderly men and women aged 60-97 years: a population-based study. PLoS One. 2013 Jul 24;8(7):e69627. doi: 10.1371/journal.pone.0069627. Print 2013. PMID 23894511
- [Background] Eendebak R, Organization WH. World report on aging and health 2015
- [Background] Kim TN, Choi KM. Sarcopenia: definition, epidemiology, and pathophysiology. J Bone Metab. 2013 May;20(1):1-10. doi: 10.11005/jbm.2013.20.1.1. Epub 2013 May 13. PMID 24524049

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT07147543/Prot_SAP_000.pdf